CLINICAL TRIAL: NCT00004489
Title: Randomized Study of Alendronate in Adult Patients With Cystic Fibrosis Related Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/14270; UNCCH-FDR001518
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-01

CONDITIONS: Osteoporosis; Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; disease-related problem/condition; genetic diseases and dysmorphic syndromes; osteoporosis; rare disease
MeSH Terms: conditions — Osteoporosis; Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Alendronate; Calcium Carbonate; Cholecalciferol

INTERVENTIONS:
Drug: alendronate sodium
Drug: calcium carbonate
Drug: cholecalciferol

SUMMARY:
OBJECTIVES: I. Determine the bioavailability and biologic effect of alendronate on bone metabolism in patients with cystic fibrosis.

II. Assess the safety and efficacy of this treatment regimen in improving osteoporosis in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study. Patients will be stratified according to sex (male vs female) and osteoporosis disease severity (mild vs severe). Patients are randomized to one of two treatment arms.

Patients undergo bioavailability assessment to confirm the ability to absorb alendronate.

Arm I: Patients receive calcium and vitamin D supplements with a placebo daily for one month.

Arm II: Patients receive calcium and vitamin D supplements with oral alendronate daily for one month.

Treatment continues if differences are seen in bone mineral density between the treatment arms.

Patients are followed for biochemical response at week 6, 12, and 52. Bone mineral density is measured at 1 year and 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of cystic fibrosis Mild to moderate lung disease
* At least one site specific (spine or femur) bone mineral density representing low bone mass or osteopenia (greater than 1 standard deviation below peak bone mass)

--Prior/Concurrent Therapy--

* Endocrine therapy: At least 3 months since prior corticosteroids

--Patient Characteristics--

* Performance status: Ambulatory
* Renal: Creatinine no greater than 3 mg/dL No renal failure
* Other: No history of esophagitis No allergies to alendronate Not pregnant Fertile female patients must use effective barrier contraception or progestin only oral contraceptives (e.g., norethindrone) Ability to comply with treatment No intestinal problems other than cystic fibrosis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 1998-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Robert Aris, Study Chair — University of North Carolina
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States